CLINICAL TRIAL: NCT02061046
Title: Impact of the CPAP on Gait in OSA Patients
Brief Title: To Study the Impact of CPAP on Gait Parameters in OSA Patients
Acronym: OSA_Gait
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Gilles Allali, Dr, University Hospital, Geneva
Other Study IDs: PRD 10-II-7
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Gait; Dual task
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- On CPAP therapy: OSA patients assessed before and after 8 weeks of CPAP therapy
  Interventions: Device: CPAP therapy

INTERVENTIONS:
Device: CPAP therapy — 8 weeks of CPAP therapy

SUMMARY:
To study the impact of CPAP therapy on gait in patients with obstructive sleep apnea syndrome.

DETAILED DESCRIPTION:
To study the impact of CPAP therapy on gait velocity and temproral gait in patients with obstructive sleep apnea syndrome using the SMTEC system. Patients will be assessed before and 8 weeks after CPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* OSA patients newly diagnosed

Exclusion Criteria:

* acute medical illness in the past months
* neurological and psychiatric diseases
* orthopaedic, rheumatologic or any sensory conditions affecting normal walking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: OSA patients without any prior treatment
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Gait parameters: gait velocity [m/s] | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Allali, MD/PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland